CLINICAL TRIAL: NCT04492878
Title: A Phase IV Open-Label Clinical Trial to Evaluate the Efficacy of Ikervis® on Clinical Parameters and Molecular/Cellular Biomarkers in Dry Eye Patients With Severe Keratitis Who Have Not Improved Despite Regular Use of Tear Substitutes Before and After Exposure to an Adverse Controlled Environment
Brief Title: Efficacy and Safety of Ikervis Under Controlled Environmental Conditions Environment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Collaborators: Santen Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOBA-ImmunEyez_011-2018
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Dry Eye; Dry Eye Syndromes; Severe Keratitis
MeSH Terms: conditions — Dry Eye Syndromes; Keratitis

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IKERVIS® (1mg/mL ciclosporin) eye drops (Experimental)
  Interventions: Drug: IKERVIS®1mg/mL

INTERVENTIONS:
Drug: IKERVIS®1mg/mL — One drop of study medication once daily in each eye at bedtime during 90 days.

SUMMARY:
The proposed study is a prospective, open-label, unicentric, phase IV clinical trial.

This study is design to find new efficacy biomarkers for IKERVIS® (1mg/mL ciclosporin) eye drops after 1 and 3 month after initiation of therapy. Additionally, this study intends to investigate whether IKERVIS® will help patients to better overcome situations of desiccating stress by exposing them to an adverse controlled environment (ACE) and analyzing both clinical and molecular parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Diagnosis of DED with Severe Keratitis who have not improved despite regular use of tear substitutes by an ophthalmologist, at least 2 months previously.
* Not stable (as defined by the two items below) under at least 2 months of constant and regular use of artificial tears (at least 4 drops a day)
* Fluorescein corneal staining ≥ 2 (Oxford scale) in both eyes.
* DEQ-5 > 6 points
* Use of at least 4 times daily of an ocular artificial tears.
* Any concomitant medication that may affect DED, ocular surface condition or vision, must have a start date at least 3 months prior to baseline and dosage is not expected to change during the study.
* Best corrected visual acuity (BCVA) of at least 0.1 logMar at 6 meters with each eye.
* Signature of written informed consent form and data protection form.

Exclusion Criteria:

* Known allergy or sensitivity to the study product(s) or its components.
* Any ocular pathology other than DED.
* History of severe ocular inflammation other than that due to DED or infection in the 6 previous months to the study inclusion.
* Any ocular surgery or trauma that may affect corneal sensitivity and/or normal tear distribution in the 6 previous months or any ocular or systemic surgery or procedure planned during the study duration that may affect the study as assessed by principal investigator.
* History of refractive surgery in the previous 18 months.
* Contact lens use in the ONE previous month to study inclusion and during the duration of the study.
* Use of any ocular topical medication for pathologies other than DED.
* Use of any other ocular topical medication for DED other than artificial tears during the last ONE (steroids) or THREE months (ciclosporine, tacrolimus) .
* Any uncontrolled severe systemic disease that may affect the eye (except for Sjögren's syndrome)
* The start date of any systemic medication that may affect DED, ocular surface condition or vision is < 3 months prior to baseline or a change in dosage is anticipated during the study.
* Occlusion of the lacrimal puncta either surgically or with plugs within one month prior to study, or anticipated use of the same during the study.
* Pregnancy or breastfeeding.
* Current enrolments in an investigational drug or device study or participation in such a study within 30 day of entry into this study at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Corneal fluoresceing staining | V1 (baseline) vs V2 (30 days of treatment); V1 (baseline) vs V3 (90 days of treatment); V2 (30 days of treatment) vs V3 (90 days of treatment)
  Significant reduction in corneal fluorescein staining

SECONDARY OUTCOMES:
Response against adverse environmental conditions | V1 (baseline) vs V2 (30 days of treatment); V1 (baseline) vs V3 (90 days of treatment)
  Significant differences in the percentage of patients suffering a worsening in clinical signs and/or symptoms following exposure to adverse environmental conditions
Molecular changes | V1 (baseline) vs V2 (30 days of treatment); V1 (baseline) vs V3 (90 days of treatment)
  Significant reduction in median expression of HLA-DR by conjunctival epithelial cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Applied Ophthalmobiology (IOBA), Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valencia-Nieto L, Pinto-Fraga J, Blanco-Vazquez M, Fernandez I, Lopez-Miguel A, Garcia-Vazquez C, Gonzalez-Garcia MJ, Enriquez-de-Salamanca A, Calonge M. Short-Term Efficacy of Ophthalmic Cyclosporine: A 0.1% Cationic Emulsion in Dry Eye Patients Assessed Under Controlled Environment. Ophthalmol Ther. 2024 May;13(5):1197-1210. doi: 10.1007/s40123-024-00906-1. Epub 2024 Mar 6. PMID 38446281